CLINICAL TRIAL: NCT06115629
Title: Open Label International Multicentre Randomised Controlled Trial of Intensive Surveillance vs. Standard Postoperative Follow-up in Patients Undergoing Surgical Resection for Oesophageal and Gastric Cancer
Brief Title: Surveillance After Resection of Oesophageal aNd Gastric Cancer (SARONG-II) Trial
Acronym: SARONG-II
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: Trinity St. James's Cancer Institute (Unknown); University of Oxford (Other); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Dr Jessie A Elliott, Clinical Lecturer, University of Dublin, Trinity College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: R&I 8335
Record Dates: First submitted 2023-10-23; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: Surveillance; Cancer recurrence; Quality of life
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Imaging surveillance (Experimental): Computed tomography scan every 6 months for 3 years postoperatively. Upper gastrointestinal endoscopy at 12 months postoperatively.
  Interventions: Other: Surveillance protocol
- Clinical surveillance (No Intervention): Clinical review every 6 months for 3 years postoperatively with further investigation according to symptoms.

INTERVENTIONS:
Other: Surveillance protocol — Imaging surveillance will entail a computed tomography scan of the chest, abdomen and pelvis, as well as clinical review, every 6 months for 36 months post surgery along with an endoscopy at 12 months post surgery.
  Arms: Imaging surveillance

SUMMARY:
Cancer of the food pipe (oesophagus) and stomach are increasingly common. Currently, most patients with cancer of the oesophagus and stomach are treated with surgery with or without additional chemotherapy or radiotherapy. In recent years there have been improvements in survival from these two cancers, due to better therapies, less invasive surgery and earlier detection. Despite these improvements, in around half of patients treated with surgery, the cancer will return, usually within the first three years.

At present there is very little evidence as to how patients who have been treated for cancer of the oesophagus or stomach should be followed up after surgery and whether different methods of follow-up could improve survival. Currently, national and international guidelines do not provide consistency in their recommendations for follow-up after surgery.

The SARONG-II study will investigate if regular radiological scans can lead to earlier detection of a cancer returning, at a stage when it may be more readily treatable. This means that participants who agree to take part will be allocated by chance to either more intensive imaging surveillance (including regular radiological scans and a camera test (endoscopy)) or clinical follow-up.

The study aims to recruit at least 952 participants in Europe over a 32-month period. Patients undergoing surgery for oesophageal or stomach cancer will be invited to participate in the study at around 4 to 8 weeks after their surgery.

(i) The imaging surveillance group will receive a review in clinic or by telephone with a member of the surgical team, and a radiological scan at 6, 12, 18, 24, 30 and 36 months after randomisation. They will also receive endoscopy at 12 months after randomisation (ii) The clinical surveillance group will receive a review in clinic or by telephone at 6, 12, 18, 24, 30 and 36 months. After this they will be either discharged to their local doctor or receive a review in clinic with a member of the surgical team every year according to local practice

The main aim of this study will be to determine whether earlier detection of cancer through more intensive follow-up results in improved survival and better quality of life for patients with oesophagus or stomach cancer. The investigators anticipate the results of the study may have significant practice-changing impact for patients undergoing follow-up after surgery for oesophagus and stomach cancer.

DETAILED DESCRIPTION:
It is an encouraging trend that the overall survival rate for oesophagogastric cancer has doubled over the last 20 years. For patients with locally advanced disease treated with curative intent, 5 year survival in the modern era approaches 50%. Relevant factors include earlier diagnosis, improvements in staging, and quality improvements in the standard modalities of surgery, chemotherapy and radiation therapy, increasingly delivered in high volume centers. When local or systemic failure occurs, where therapeutic nihilism may have once prevailed, a menu of therapeutic options can now be considered, such as immunotherapy, salvage locoregional surgery, resection of oligometastatic disease, brachytherapy, radiofrequency ablation (RFA) and stereotactic radiation therapy.

In the context of this changing landscape and expanded armamentarium, a key question, as yet unresolved, is how patients treated with curative intent should be optimally followed-up. The options include an intensive imaging surveillance approach using clinical assessment, cross-sectional imaging, and endoscopy, or one purely based on symptomatic follow-up to trigger further investigation.

The debate for oesophagogastric cancer is limited by a paucity of evidence. This may reflect both a lack of attention to this topic in research, with no RCTs, and relatively poor quality cohort and observational studies with considerable heterogeneity. The approach to surveillance varies considerably internationally. In Japan, a nationwide survey reported that that high intensity surveillance was common, with endoscopic surveillance utilized in over 80% of patients, in contrast to approximately 6% in Australia and New Zealand. In Europe, the European Registration of Cancer Care (EURECCA) Upper Gastrointestinal group reported a brief summary from 10 Centers, and highlighted substantial differences in elements of surveillance, in particular of cross-sectional imaging, which was sought in just 40% of patients. Guidelines also vary, for instance the European Society for Medical Oncology guidelines currently state, "With the exception of endoscopic or operative salvage after initial non-operative management, there is no evidence that regular follow-up has an impact on survival outcomes", while the UK NICE guidelines state, "for people without symptoms or evidence of residual disease after treatment for oesophagogastric cancer with curative intent, do not offer routine clinical follow-up or radiological surveillance solely for the detection of recurrent disease".

It is clear that research is urgently required on this important topic that will inform everyday practice and future guidelines. In this context, a European collaborative multicenter study was established with the primary objective of assessing the current situation in specialist centers internationally and its impact on survival and quality of life.

In this study, the investigators first surveyed 27 European centres, and identified marked variation in surveillance practices, with only 37% of centres providing routine radiologic surveillance for detection of recurrence, and only 19% undertaking routine surveillance endoscopy. The investigators then undertook a European multicentre cohort study, which included 4682 patients. At median follow-up 60 months, 47.5% developed recurrence, oligometastatic in 39%. Intensive surveillance, defined as a computed tomography scan undertaken at least annually for three years after surgery, was associated with reduced symptomatic recurrence and increased tumor-directed therapy. On multivariable analysis, no overall survival benefit was observed among all patients (HR1.01 [0.89-1.13]), but overall survival was improved following intensive surveillance for those who underwent surgery alone and those with lower pathological (y)pT stages. Intensive surveillance was associated with similar overall HRQL. This study established that there is widespread heterogeneity in surveillance protocols in Europe, and the vast majority of centres agreed there is a need for an RCT examining this issue.

The SARONG-II study is an international multicentre, open-label, two-arm, parallel design, superiority randomised controlled trial. 952 patients (476 in each of two trial arms) will be recruited from approximately 14 sites in Europe. Participants will be randomised to either imaging surveillance every 6 months for 36 months and an endoscopy at 12 months postrandomisation or clinical follow-up for 36 months.

Primary Outcome Measure:

All-cause mortality defined as death from any cause. Participants who have not been observed to die during the course of the study will have their survival time censored at their last known follow-up date.

Secondary Outcome Measures:

1. a) Disease-specific mortality, defined as known oesophageal or gastric cancer recurrence at the time of death.

   b) Pattern of tumour recurrence, defined as the incidence of loco-regional or distant recurrence.

   c) Treatment of tumour recurrence, ie. the requirement for chemotherapy, surgery, immunotherapy, radiotherapy, chemoradiotherapy, best supportive care or other as determined by the clinical team at the treating site.

   d) Rates of oligometastatic (one site) tumour recurrence. e) Rates of multi-metastatic (several sites) tumour recurrence.
2. HRQoL, including anxiety or depression and worry of cancer returning as measured by the following validated questionnaires: EQ- 5D-5L, EORTC QLQ-C30 and QLQ-OG25 and Cancer Worry Scale (CWS).
3. Incremental cost per quality adjusted life year (QALY)

ELIGIBILITY:
A patient will be eligible for inclusion in this study if all of the following criteria apply:

1. Has undergone surgical resection for curatively intended treatment of oesophageal or gastric cancer (adenocarcinoma and squamous cell carcinoma) with or without neoadjuvant/adjuvant chemotherapy or radiotherapy or immunotherapy (or in combination).
2. Aged 18 years or over
3. Willing and able to give informed consent

A patient with not be eligible for the trial if any of the following apply:

1. Other cancer(s) undergoing treatment or surveillance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 952 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 36 months post randomisation
  All-cause mortality defined as death from any cause. Participants who have not been observed to die during the course of the study will have their survival time censored at their last known follow-up date.

SECONDARY OUTCOMES:
Disease-specific mortality | 36 months post randomisation
  Disease-specific mortality, defined as known oesophageal or gastric cancer recurrence at the time of death.
Pattern of recurrence | 36 months post randomisation
  Pattern of tumour recurrence, defined as the incidence of loco-regional or distant recurrence.
Treatment of recurrence | 36 months post randomisation
  Treatment of tumour recurrence, ie. the requirement for chemotherapy, surgery, immunotherapy, radiotherapy, chemoradiotherapy, best supportive care or other as determined by the clinical team at the treating site.
Oligometastatic recurrence as determined using the OligoMetastatic Esophagogastric Cancer (OMEC) classification system | 36 months post randomisation
  Rates of oligometastatic tumour recurrence
Multimetastatic recurrence | 36 months post randomisation
  Rates of multi-metastatic (several sites) tumour recurrence
Overall quality of life as determined by the global health status using the European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire C30 | 36 months post randomisation
  Using European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire C30, reported as a linear transformed outcome ranging from 0-100.
Cost effectiveness as determined by incremental cost per quality adjusted life year | 36 months post randomisation
  Incremental cost per quality adjusted life year (QALY) determined using the 5-level EQ-5D version (EQ-5D-5L) as well as healthcare utilisation costs measured in Euro.
Fear of cancer recurrence as determined by the cancer worry scale score | 36 months post randomisation
  Measured from 1-4

CONTACTS AND LOCATIONS:
Overall Officials: Jessie A Elliott, PhD FRCS, Principal Investigator — Trinity St. James's Cancer Institute
Locations (13):
- University Hospital Cologne, Cologne, Germany
- Ireland (3):
  - Mercy University Hospital, Cork
  - Trinity St. James's Cancer Institute, Dublin
  - Galway University Hospital, Galway
- Fondazione Policlinico Universitario Agostino Gemelli, Roma, Italy
- Norway (3):
  - Oslo University Hospital, Oslo
  - University Hospital of Northern Norway, Tromsø
  - St. Olav University Hospital, Trondheim
- Sweden (5):
  - Linköping University Hospital, Linköping
  - Skåne University Hospital, Lund
  - Örebro University Hospital, Örebro
  - Karolinska Institutet, Stockholm
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Elliott JA, Klevebro F, Mantziari S, Markar SR, Goense L, Johar A, Lagergren P, Zaninotto G, van Hillegersberg R, van Berge Henegouwen MI, Schafer M, Nilsson M, Hanna GB, Reynolds JV; ENSURE Study Group. Neoadjuvant Chemoradiotherapy Versus Chemotherapy for the Treatment of Locally Advanced Esophageal Adenocarcinoma in the European Multicenter ENSURE Study. Ann Surg. 2023 Nov 1;278(5):692-700. doi: 10.1097/SLA.0000000000006018. Epub 2023 Jul 20. PMID 37470379
- [Background] Gujjuri RR, Clarke JM, Elliott JA, Rahman SA, Reynolds JV, Hanna GB, Markar SR; ENSURE Group Study. Predicting long-term survival and time-to-recurrence after esophagectomy in patients with esophageal cancer - Development and validation of a multivariate prediction model. Ann Surg. 2023 Jun;277(6):971-978. doi: 10.1097/SLA.0000000000005538. Epub 2022 Jul 15. No abstract available. PMID 37193219
- [Background] Elliott JA, Markar SR, Klevebro F, Johar A, Goense L, Lagergren P, Zaninotto G, van Hillegersberg R, van Berge Henegouwen MI, Nilsson M, Hanna GB, Reynolds JV; ENSURE Study Group. An International Multicenter Study Exploring Whether Surveillance After Esophageal Cancer Surgery Impacts Oncological and Quality of Life Outcomes (ENSURE). Ann Surg. 2023 May 1;277(5):e1035-e1044. doi: 10.1097/SLA.0000000000005378. Epub 2022 Jan 27. PMID 35129466
- [Background] Chidambaram S, Sounderajah V, Maynard N, Underwood T, Markar SR. Evaluation of postoperative surveillance strategies for esophago-gastric cancers in the UK and Ireland. Dis Esophagus. 2022 Feb 11;35(2):doab057. doi: 10.1093/dote/doab057. PMID 34426840
- [Background] Chidambaram S, Sounderajah V, Maynard N, Markar SR. Evaluation of post-operative surveillance strategies for esophageal and gastric cancers: a systematic review and meta-analysis. Dis Esophagus. 2022 Dec 14;35(12):doac034. doi: 10.1093/dote/doac034. PMID 35788834